CLINICAL TRIAL: NCT04757792
Title: Back to the Traditional: Anti-COX Drugs Can Improve the Outcome of COVID-19 Patients Admitted to ICU
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Collaborators: Tanta University (Other); Cairo University (Other)
Responsible Party: Principal Investigator, Adel F. Alkholy, Professor of Medical Biochemistry, Benha University
Other Study IDs: RC1-2-2021
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: COVID-19 Disease
Keywords: COVID-19; NSAID; Aspirin; Mortality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- No NSAID: included patients who did not receive NSAID prior to having COVID-19 disease
  Interventions: Other: File inquiry
- Apsirin: included patients who received acetylsalicylic acid (ASA) prior to having COVID-19 disease
  Interventions: Other: File inquiry
- Celecoxib: included patients who received celecoxib (CEL) prior to having COVID-19 disease
  Interventions: Other: File inquiry
- Miscellaneous: included patients who received miscellaneous NSAID other than ASA or CEL prior to having COVID-19 disease
  Interventions: Other: File inquiry

INTERVENTIONS:
Other: File inquiry — Data extraction out of file registry
  Other Names: No interventions

SUMMARY:
Retrospective multicenter study to evaluate the data of COVID-19 patients who were admitted to university hospitals in relation to their recent administration or maintenance on non-steroidal anti-inflammatory drugs (NSAID) prior to have COVID-19 disease and to analyze it in relation to outcome of these patients.

DETAILED DESCRIPTION:
The data contained in hospital registry were collected, categorized into demographic, previous medical history, the use of NSAID as maintenance therapy or its recent administration before diagnosis of COVID-19 disease, presenting manifestations, laboratory and CT findings, applied therapies or interventions. Outcomes will be categorized as survival and non-survival outcome. Survivors will be subdivided as complete recovery or recovery with getting new morbidities. Mortality was subdivided as total hospital and ICU mortality. Data will be statistically analyzed in relation to outcomes

ELIGIBILITY:
Inclusion Criteria:

* assured diagnosis of COVID-19 by RT-PCR

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with diagnosis of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 6 months
  number of patients who were died secondary to COVID-19 disease or its complications

CONTACTS AND LOCATIONS:
Overall Officials: Adel Alkholy, Prof, Principal Investigator — Faculty of medicine, Banha University, Egypt
Locations (1):
- Faculty of Medicine, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Protocol data will be available on request
Supporting Information: Study Protocol
Time Frame: After publishing
Access Criteria: email